CLINICAL TRIAL: NCT01907100
Title: LUME-Meso: Double Blind, Randomised, Multicentre, Phase II/III Study of Nintedanib in Combination With Pemetrexed / Cisplatin Followed by Continuing Nintedanib Monotherapy Versus Placebo in Combination With Pemetrexed / Cisplatin Followed by Continuing Placebo Monotherapy for the Treatment of Patients With Unresectable Malignant Pleural Mesothelioma
Brief Title: Nintedanib (BIBF 1120) in Mesothelioma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.93; 2012-005201-48 (EudraCT Number)
Record Dates: First submitted 2013-07-22; First posted 2013-07-24 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — nintedanib; Pemetrexed; Cisplatin

ARMS (2):
- Placebo + pemetrexed/cisplatin (Placebo Comparator): Placebo controlled arm
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Placebo
- Nintedanib 200mg + pemetrexed/cisplatin (Experimental): Experimental arm
  Interventions: Drug: Nintedanib; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Nintedanib — triple kinase inhibitor; 200mg starting dose
  Arms: Nintedanib 200mg + pemetrexed/cisplatin
Drug: Pemetrexed — backbone chemo
  Arms: Placebo + pemetrexed/cisplatin
Drug: Cisplatin — backbone chemo
  Arms: Nintedanib 200mg + pemetrexed/cisplatin
Drug: Cisplatin — backbone chemo
  Arms: Placebo + pemetrexed/cisplatin
Drug: Pemetrexed — backbone chemo
  Arms: Nintedanib 200mg + pemetrexed/cisplatin
Drug: Placebo — Nintedanib matching placebo
  Arms: Placebo + pemetrexed/cisplatin

SUMMARY:
This is a phase II/III confirmatory study designed to evaluate the safety and efficacy of nintedanib (BIBF 1120) in combination + (pemetrexed / cisplatin) followed by nintedanib (BIBF 1120) versus placebo + pemetrexed / cisplatin followed by placebo for the treatment of patients with unresectable malignant pleural mesothelioma.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed malignant pleural mesothelioma (MPM) (Epithelioid or biphasic subtype for Phase II patients; epithelioid subtype only for Phase III patients)
* Life expectancy of at least 3 months in the opinion of the investigator
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Measurable disease according to modified RECIST (Response Evaluation Criteria In Solid Tumours) criteria

Exclusion criteria:

* Previous systemic chemotherapy for MPM
* Prior treatment with nintedanib or any other prior line of therapy
* Phase II patients with sarcomatoid subtype MPM or Phase III patients with biphasic or sarcomatoid subtype MPM
* Patients with symptomatic neuropathy
* Radiotherapy (except extremities) within 3 months prior to baseline imaging
* Active brain metastases (e.g. stable for < 4 weeks)
* Radiographic evidence of cavitary or necrotic tumours or local invasion of major blood vessels by MPM
* Significant cardiovascular diseases
* Inadequate hematologic, renal, or hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (123):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology-San Antonio Northeast, San Antonio, Texas
  - Cancer Care Northwest Centers, PS, Spokane Valley, Washington
- Argentina (3):
  - Sanatorio Güemes, Ciudad Autónoma de Bs As
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autónoma de Bs As
  - Clínica Universitaria Reina Fabiola, Córdoba
- Australia (10):
  - Northern Cancer Institute, St Leonards, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Peninsula Haematology & Oncology, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - Border Onclogy Research, Wodonga, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Perth Oncology, Perth, Western Australia
- Austria (3):
  - LKH Leoben, Leoben
  - AKH - Medical University of Vienna, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (5):
  - Brussels - UNIV Saint-Luc, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
  - AZ Sint-Maarten, Mechelen
- Canada (4):
  - QEII Health Sciences Centre (Dalhousie University), Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - IUCPQ (Laval University), Québec
- Chile (2):
  - Centro Internacional de Estudios Clínicos - CIEC, Recoleta
  - Orlandi Oncologia, Vitacura
- University Clinic for Pulmonary Diseases, Zagreb, Croatia
- Czechia (2):
  - University Hospital Brno, Brno
  - University Hospital Olomouc, Olomouc
- Rigshospitalet, København, Onkologisk afdeling, Købenahvn Ø, Denmark
- Egypt (4):
  - Clinical Research Center Alexandria, Alexandria
  - Medical Research Institute, Alexandria
  - National Cancer Institute, Cairo University, Cairo
  - Nasser Institute, Cairo
- France (9):
  - CLI Bordeaux Nord Aquitaine, Bordeaux
  - HOP Morvan, Brest
  - HOP Côte de Nacre, Caen
  - HOP Calmette, Lille
  - HOP Nord, Marseille
  - HOP Lyon Sud, Pierre-Bénite
  - HOP HIA Saint-Anne, Toulon
  - HOP Larrey, Toulouse
  - INS Gustave Roussy, Villejuif
- Germany (7):
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Klinik Schillerhöhe GmbH, Gerlingen
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinik, Löwenstein, Löwenstein
- Israel (3):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Centro di riferimento Oncologico, Aviano (PN)
  - Humanitas Gavazzeni, Bergamo
  - Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano (TO)
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (8):
  - University Hospital of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Hyogo Prefectural Amagasaki General Medical Center, Hyogo, Amagasaki
  - Hyogo College of Medicine Hospital, Hyogo, Nishinomiya
  - Yokosuka Kyosai Hospital, Kanagawa , Yokosuka
  - Japan Labour Health and Safety Organization Okayama Rosai Hospital, Okayama, Okayama
  - Kindai University Hospital, Osaka, OsakaSayama
  - Otemae Hospital, Osaka, Osaka
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
- Mexico (3):
  - Centro Oncologico de Chihuahua, Chihuahua City
  - Instituto Nacional de Cancerologia, México
  - Centro Oncologico Estatal ISSEMYM, Toluca
- Netherlands (3):
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Medisch Centrum, Heerlen
  - Erasmus Medisch Centrum, Rotterdam
- Norway (2):
  - Oslo Universitetssykehus HF, Radiumhospitalet, Oslo
  - St. Olavs Hospital, Universitetssykehuset i Trondheim, Trondheim
- Poland (4):
  - University Clinical Center, Gdansk, Gdansk
  - Clin.Hosp.Med.Univ.Marcinkowski in Poznan, Poznan
  - Greater PL Cent.Pulmo.&Thor.Surg.Eugenia&Janusz Zeyland, Poznan
  - Onco.Cent. - Instit. of Maria Sklodowskiej-Curie, Warsaw
- Portugal (2):
  - Centro Hospitalar Lisboa Norte Hospital Pulido Valente, Lisbon
  - Hospital CUF Porto, Porto
- Russia (6):
  - St.Budg.Heal.Inst."Chelyabinsk Reg.Clin.Cen.Onc&Nucl.Med", Chelyabinsk
  - St.Auton.Heal.Inst."Rep.Clin.Onc.Disp.of MoH of Rep. Tatarstan", Kazan'
  - FSBI "N.N Blokhin Med.Res.Cent.Onc."MoH of RF, Moscow
  - 1stPavlov St.Med.Univ.St.-Petersburg Res.Inst., Saint Petersburg
  - FSBI "N.N. Petrov National Medical Research Center of Oncology" of MoH of RF, Saint Petersburg
  - SBI HC-Rep.Clin.Onc.Disp.MoH.Rep.Bashkortostan, Ufa
- Wilgers Oncology Centre, Pretoria, South Africa
- Spain (9):
  - Hospital Universitario de Cruces, Barakaldo (Vizcaya)
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Donostia, Donostia (Gipuzkoa)
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Ramón y Cajal, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico de Valencia, Valencia
- Sweden (5):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Universitetssjukhuset, Linköping, Linköping
  - Skånes universitetssjukhus, Lund, Lund
  - Karolinska Univ. sjukhuset, Stockholm
  - Akademiska sjukhuset, Uppsala
- Turkey (Türkiye) (3):
  - Eskisehir Osmangazi Üni. Sag. Uygulama ve Arastirma Has., Eskişehir
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Dr.Suat Seren EAH, Izmir
- United Kingdom (7):
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Guy's Hospital, London
  - The Royal Marsden Hospital, London
  - The Royal Marsden Hospital, Sutton
  - Wythenshawe Hospital, Wythenshawe

REFERENCES:
- [Derived] Scagliotti GV, Gaafar R, Nowak AK, Nakano T, van Meerbeeck J, Popat S, Vogelzang NJ, Grosso F, Aboelhassan R, Jakopovic M, Ceresoli GL, Taylor P, Orlandi F, Fennell DA, Novello S, Scherpereel A, Kuribayashi K, Cedres S, Sorensen JB, Pavlakis N, Reck M, Velema D, von Wangenheim U, Kim M, Barrueco J, Tsao AS. Nintedanib in combination with pemetrexed and cisplatin for chemotherapy-naive patients with advanced malignant pleural mesothelioma (LUME-Meso): a double-blind, randomised, placebo-controlled phase 3 trial. Lancet Respir Med. 2019 Jul;7(7):569-580. doi: 10.1016/S2213-2600(19)30139-0. Epub 2019 May 15. PMID 31103412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were initially treated with combination therapy consisting of nintedanib or placebo plus standard chemotherapy (pemetrexed/cisplatin), for a maximum of 6 cycles of 21 days duration. After completion of combination therapy, patients who had not progressed continued with nintedanib or placebo monotherapy.
Pre-assignment Details: All participants were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the participants) met all implemented inclusion/exclusion criteria. Participants were not to be entered to trial if any of the specific entry criteria was violated.
  PD: Progressive Disease
Groups:
- Placebo_Phase II: Phase II part:
  Nintedanib matching placebo 200 mg twice daily (b.i.d.) on Day 2 to 21 of each 21-day treatment course administered orally in the form of a soft gelatin capsule (100 mg or 150 mg capsules) plus standard Pemetrexed 500 mg/m2 (100 mg or 500 mg vials) and Cisplatin 75 mg/m2 (50 mL of 1 mg/ml solution) on Day 1 of each 21-day treatment course administered intravenously. If required, the dose of placebo could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
- Nintedanib_Phase II: Phase II part: Nintedanib 200 mg twice daily (b.i.d.) on Day 2 to 21 of each 21-day treatment course administered orally in the form of a soft gelatin capsule (100 mg or 150 mg capsules) plus standard Pemetrexed 500 mg/m2 (100 mg or 500 mg vials) and Cisplatin 75 mg/m2 (50 mL of 1 mg/ml solution) on Day 1 of each 21-day treatment course administered intravenously. If required, the dose of Nintedanib could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
- Placebo_Phase III: Phase III part: Nintedanib matching Placebo 200 mg twice daily (b.i.d.) on Day 2 to 21 of each 21-day treatment course administered orally in the form of a soft gelatin capsule (100 mg or 150 mg capsules) plus standard Pemetrexed 500 mg/m2 (100 mg or 500 mg vials) and Cisplatin 75 mg/m2 (50 mL of 1 mg/ml solution) on Day 1 of each 21-day treatment course administered intravenously. If required, the dose of placebo could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
- Nintedanib_Phase III: Phase III part: Nintedanib 200 mg twice daily (b.i.d.) on Day 2 to 21 of each 21-day treatment course administered orally in the form of a soft gelatin capsule (100 mg or 150 mg capsules) plus standard Pemetrexed 500 mg/m2 (100 mg or 500 mg vials) and Cisplatin 75 mg/m2 (50 mL of 1 mg/ml solution) on Day 1 of each 21-day treatment course administered intravenously. If required, the dose of Nintedanib could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
Period: Overall Study
Arm/Group | Placebo_Phase II | Nintedanib_Phase II | Placebo_Phase III | Nintedanib_Phase III
Started | 43 | 44 | 229 | 229
Treated Patients | 41 | 44 | 228 | 227
Completed (On treatment or completed according to protocol at the time of analysis) | 1 | 4 | 82 | 83
Not Completed | 42 | 40 | 147 | 146
Not completed — PD based on modified RECIST criteria | 31 | 32 | 95 | 92
Not completed — Withdrawal by Subject | 2 | 5 | 10 | 13
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Not treated | 2 | 0 | 1 | 2
Not completed — Other than reasons specified | 1 | 0 | 10 | 6
Not completed — Adverse event (AE) | 6 | 3 | 22 | 23
Not completed — Worsening/AE underlying cancer disease | 0 | 0 | 8 | 8

BASELINE CHARACTERISTICS:
Population: Randomised Set: This patient set included all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo_Phase II | Nintedanib_Phase II | Placebo_Phase III | Nintedanib_Phase III | Total
Number analyzed (Participants) | 43 | 44 | 229 | 229 | 545
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (7.6) | 66.4 (8.6) | 64.3 (8.9) | 63.6 (9.5) | 64.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 60 | 64 | 142
  Male | 35 | 34 | 169 | 165 | 403
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data were not collected from any participant
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was only collected where allowed by local law.
  Participants
    American Indian or Alaska Native | 0 | 0 | 14 | 12 | 26
    Asian | 0 | 0 | 16 | 14 | 30
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 2 | 2
    White | 38 | 38 | 180 | 185 | 441
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 5 | 6 | 19 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: This outcome measure presents progression-free survival. Disease progression was defined according to the modified Response Evaluation Criteria in Solid Tumours (RECIST) criteria. Progression-free survival time was calculated as the duration from the date of randomization to the date of disease progression or death, whichever occurred first. For patients with known date of progression (or death): PFS (days) = min (date of progression, date of death) - date of randomization + 1 day. For patients without progression or death, PFS was censored at the last imaging date that showed no disease progression: PFS (days, censored) = date of last imaging showing no progression - date randomization + 1 day.
Time Frame: From randomization until the earliest of disease progression, death or (Phase II: cut-off date of 4-March-2016; up to 889 days) (Phase III: cut-off date of 16-March-2018; up to 31 months)
Population: Randomised Set: This patient set included all randomized patients.
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- Placebo: Nintedanib matching Placebo 200 mg twice daily (b.i.d.) on Day 2 to 21 of each 21-day treatment course administered orally in the form of a soft gelatin capsule (100 mg or 150 mg capsules) plus standard Pemetrexed 500 mg/m2 (100 mg or 500 mg vials) and Cisplatin 75 mg/m2 (50 mL of 1 mg/ml solution) on Day 1 of each 21-day treatment course administered intravenously. If required, the dose of placebo could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
- Nintedanib: Nintedanib 200 mg twice daily (b.i.d.) on Day 2 to 21 of each 21-day treatment course administered orally in the form of a soft gelatin capsule (100 mg or 150 mg capsules) plus standard Pemetrexed 500 mg/m2 (100 mg or 500 mg vials) and Cisplatin 75 mg/m2 (50 mL of 1 mg/ml solution) on Day 1 of each 21-day treatment course administered intravenously. If required, the dose of Nintedanib could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 272 | 273
Months
  Phase II: number analyzed (Participants) | 43 | 44
  Phase II | 5.72 [5.19 to 8.18] | 9.36 [5.55 to 12.65]
  Phase III: number analyzed (Participants) | 229 | 229
  Phase III | 6.97 [5.42 to 9.00] | 6.77 [5.36 to 9.07]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Phase II Part; Test type: Other; p = 0.0174, Proportional hazards mode; Hazard Ratio (HR) = 0.555, 95% CI 2-sided [0.340 to 0.907] — Hazard ratio, confidence interval and p-value obtained from proportional hazards model stratified by tumour histology (epithelioid vs. biphasic)
Statistical Analysis 2: Comparison: Placebo vs Nintedanib; Phase III part: A Cox proportional hazards model was fitted to estimate hazard ratios (HRs) and corresponding 95% confidence intervals (CIs) for the comparison of treatment arms (Nintedanib vs Placebo). If the hazard ratio is below 1 then it favours nintedanib; Test type: Other; p = 0.5430, Proportional hazards model — one-sided p-value; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.79 to 1.30] — Hazard ratio, confidence interval and p-value obtained from a non-stratified proportional hazards model

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the duration of time from randomization to time of death.
  This is the key secondary endpoint of the trial.
Time Frame: as for outcome 1
Population: Randomised Set: This patient set included all randomized patients.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 272 | 273
Months
  Phase II: number analyzed (Participants) | 43 | 44
  Phase II | 14.46 [10.41 to NA] — The 75th percentile was not reached because of insufficient number of patients with OS event thus not calculated. | 18.30 [10.91 to NA] — The 75th percentile was not reached because of insufficient number of patients with OS event thus not calculated.
  Phase III: number analyzed (Participants) | 229 | 229
  Phase III | 16.07 [9.66 to 19.29] | 14.36 [9.13 to 18.69]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Phase II; Test type: Other; p = 0.4132, Proportional hazards mode; Hazard Ratio (HR) = 0.782, 95% CI 2-sided [0.433 to 1.412] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Nintedanib; Phase III: A Cox proportional hazards model was fitted to estimate hazard ratios (HRs) and corresponding 95% confidence intervals (CIs) for the comparison of treatment arms (Nintedanib vs Placebo). If the hazard ratio is below 1 then it favours nintedanib; Test type: Other; p = 0.7306, Proportional hazards model — one-sided p-value; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.79 to 1.58] — Hazard ratio, confidence interval and p-value obtained from a non-stratified proportional hazards model

3. Secondary Outcome: Objective Response According to Modified RECIST- Investigator Assessment
Description: Objective response (best overall tumour response of confirmed complete response [CR] or confirmed partial response [PR]).
  Complete Response: disappearance of all target lesions Partial Response: at least a 30 % decrease in the total tumour measurement of target lesions, taking as reference the baseline total tumour measurement.
  Percentage of Patients with confirmed objective response is presented. This endpoint was only evaluated for Phase III part.
Time Frame: Tumour imaging was to be performed every 6 weeks until disease progression, death or start of subsequent anti-cancer therapy, whichever occurred earlier; up to 54 months
Population: Randomised Set: This patient set included all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 229 | 229
Percentage of participants | 42.8 [36.3 to 49.5] | 45.0 [38.4 to 51.7]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Test type: Other; p = 0.3189, Regression, Logistic — one-sided p-value; Odds ratio and one-sided p-value are obtained from an un-adjusted logistic regression model (Nintedanib vs Placebo); Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.76 to 1.58] — Odds ratio above 1 favours nintedanib; Exact 95% CI by Clopper and Pearson

4. Secondary Outcome: Disease Control According to Modified RECIST- Investigator Assessment
Description: Disease control (best overall response of confirmed CR or PR, or Stable Disease (SD) that lasted ≥36 days) according to modified RECIST.
  Percentage of Patients with Disease control is presented. This endpoint was only evaluated for Phase III part.
Time Frame: as for outcome 3
Population: Randomised Set: This patient set included all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 229 | 229
Percentage of participants | 92.6 [88.4 to 95.6] | 90.8 [86.3 to 94.2]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Test type: Other; p = 0.7512, Regression, Logistic — one-sided p-value; Odds ratio and one-sided p-value are obtained from an un-adjusted logistic regression model (Nintedanib vs Placebo); Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.40 to 1.55] — Odds ratio above 1 favours nintedanib

ADVERSE EVENTS:
Time Frame: SAE & Non SAE: From first dose until 28 days (Phase II) or 30 days (Phase III) after last dose, up to approximately (approx.) 30 months in Phase II and approx. 32 months in Phase III. All-cause mortality: From randomization until end of follow-up, up to approx. 30 months in Phase II and approx. 32 months in Phase III
Description: All-cause mortality numbers are based on randomized set whereas Serious Adverse Events (SAE) and non-SAE are based on treated set.
Arm/Group | Placebo_Phase II | Nintedanib_Phase II | Placebo_Phase III | Nintedanib_Phase III
All-Cause Mortality (participants affected / at risk) | 25/43 | 22/44 | 63/229 | 64/229
Serious Adverse Events (participants affected / at risk) | 17/41 | 16/44 | 89/228 | 99/227
Other Adverse Events (participants affected / at risk) | 41/41 | 44/44 | 219/228 | 218/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo_Phase II (N=41) | Nintedanib_Phase II (N=44) | Placebo_Phase III (N=228) | Nintedanib_Phase III (N=227)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 8 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 7 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 7 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 4 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 8 | 6
Asthenia (General disorders) | 0 | 1 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 3 | 2
General physical health deterioration (General disorders) | 1 | 0 | 2 | 4
Pyrexia (General disorders) | 2 | 3 | 10 | 4
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 4
Sepsis (Infections and infestations) | 1 | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 3
Fibrin D dimer increased (Investigations) | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 8 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 7 | 13
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 2 | 3
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 5 | 5
Death (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 3 | 2
Pain (General disorders) | 0 | 0 | 2 | 1
Performance status decreased (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 3
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Oral bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 4 | 6
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 3
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 5 | 9
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 4 | 0
Erosive balanitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 1 | 2
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1
Subclavian artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphatic obstruction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo_Phase II (N=41) | Nintedanib_Phase II (N=44) | Placebo_Phase III (N=228) | Nintedanib_Phase III (N=227)
Anaemia (Blood and lymphatic system disorders) | 9 | 16 | 94 | 76
Leukopenia (Blood and lymphatic system disorders) | 5 | 2 | 28 | 20
Neutropenia (Blood and lymphatic system disorders) | 9 | 22 | 82 | 83
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 7 | 18 | 13
Tinnitus (Ear and labyrinth disorders) | 9 | 4 | 24 | 15
Dry eye (Eye disorders) | 3 | 0 | 4 | 12
Lacrimation increased (Eye disorders) | 4 | 7 | 18 | 14
Abdominal pain (Gastrointestinal disorders) | 3 | 11 | 10 | 24
Abdominal pain upper (Gastrointestinal disorders) | 3 | 9 | 11 | 14
Constipation (Gastrointestinal disorders) | 19 | 17 | 73 | 60
Diarrhoea (Gastrointestinal disorders) | 15 | 29 | 47 | 118
Dyspepsia (Gastrointestinal disorders) | 11 | 3 | 20 | 14
Nausea (Gastrointestinal disorders) | 34 | 37 | 134 | 156
Stomatitis (Gastrointestinal disorders) | 5 | 3 | 16 | 22
Vomiting (Gastrointestinal disorders) | 20 | 24 | 66 | 96
Asthenia (General disorders) | 12 | 14 | 46 | 53
Chest pain (General disorders) | 9 | 7 | 23 | 23
Fatigue (General disorders) | 15 | 18 | 62 | 60
Mucosal inflammation (General disorders) | 4 | 7 | 22 | 16
Oedema peripheral (General disorders) | 5 | 5 | 16 | 16
Pyrexia (General disorders) | 4 | 7 | 22 | 17
Nasopharyngitis (Infections and infestations) | 1 | 4 | 12 | 9
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 6 | 16
Urinary tract infection (Infections and infestations) | 5 | 0 | 14 | 12
Alanine aminotransferase increased (Investigations) | 1 | 17 | 10 | 35
Aspartate aminotransferase increased (Investigations) | 1 | 13 | 9 | 32
Blood creatinine increased (Investigations) | 4 | 6 | 26 | 21
Blood magnesium decreased (Investigations) | 6 | 10 | 12 | 17
Gamma-glutamyltransferase increased (Investigations) | 1 | 10 | 13 | 25
Neutrophil count decreased (Investigations) | 3 | 8 | 26 | 28
Weight decreased (Investigations) | 9 | 8 | 23 | 20
Decreased appetite (Metabolism and nutrition disorders) | 16 | 17 | 66 | 66
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 13 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 13 | 20 | 20
Dizziness (Nervous system disorders) | 5 | 3 | 18 | 14
Dysgeusia (Nervous system disorders) | 11 | 11 | 27 | 27
Headache (Nervous system disorders) | 4 | 5 | 23 | 16
Lethargy (Nervous system disorders) | 13 | 6 | 5 | 13
Neuropathy peripheral (Nervous system disorders) | 6 | 9 | 18 | 13
Paraesthesia (Nervous system disorders) | 4 | 4 | 19 | 20
Insomnia (Psychiatric disorders) | 4 | 8 | 12 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 15 | 33 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 26 | 34
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 20 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 6 | 8 | 12
Rash (Skin and subcutaneous tissue disorders) | 7 | 11 | 23 | 22
Hypertension (Vascular disorders) | 6 | 6 | 21 | 26
White blood cell count decreased (Investigations) | 1 | 2 | 15 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 15 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 14 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 13 | 20
Hypoacusis (Ear and labyrinth disorders) | 1 | 4 | 4 | 7
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 3 | 11 | 7
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 2 | 5
Conjunctivitis (Infections and infestations) | 2 | 4 | 11 | 11
Influenza (Infections and infestations) | 2 | 3 | 4 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 9 | 6 | 7
Blood glucose increased (Investigations) | 1 | 5 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 3 | 1 | 1
Blood potassium decreased (Investigations) | 2 | 4 | 0 | 0
Blood urea increased (Investigations) | 3 | 8 | 10 | 9
Haemoglobin decreased (Investigations) | 2 | 4 | 2 | 1
Platelet count decreased (Investigations) | 4 | 8 | 7 | 9
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 8 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 9 | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 10 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 11 | 5
Neurotoxicity (Nervous system disorders) | 3 | 1 | 4 | 8
Depression (Psychiatric disorders) | 3 | 1 | 2 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 4 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 7 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 10 | 3

LIMITATIONS AND CAVEATS:
In accordance with the specifications in the protocol, the trial was discontinued prematurely after the primary PFS analysis not because of any safety concerns but rather due to failure to meet the efficacy target.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT01907100/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT01907100/SAP_001.pdf